CLINICAL TRIAL: NCT06614478
Title: Frailty in Hip Fracture Patients Treated With Surgery; the Role of Simple Inflammatory Biomarkers. An Observational Study
Brief Title: Frailty, Hip Fractures and Inflammatory Biomarkers
Status: Recruiting | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Chair, Professor of Anaesthesiology, University of Thessaly
Other Study IDs: Frailty and hip fractures
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Frailty; Hip Fracture; Inflammatory Biomarkers
MeSH Terms: conditions — Frailty; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hip fracture patients treated with surgery: Hip fracture patients treated with surgery. Frailty will be categorized based on the validated Groningen Frailty Indicator (GFI)

SUMMARY:
We ought to investigate if hip fracture patients suffering from frailty have higher inflammatory burden according to simple inflammatory biomarkers.

DETAILED DESCRIPTION:
Frailty (F) is a prevalent syndrome among elderly patient with hip fractures (HF) and has been linked to poor prognosis. Inflammatory biomarkers have been used as prognostic indexes in patients with HF. We ought to investigate if hip fracture patients suffering from frailty have higher inflammatory burden according to simple inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* age >65 years, ASA PS I-III, non- institutionalized, able to communicate patients

Exclusion Criteria:

* Patients with severe cognitive dysfunction, those treated conservatively, those with pathological fractures and patients who refused to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: hip fracture patients treated with surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Frailty status | preoperatively
  Frailty will be categorized based on the validated Groningen Frailty Indicator (GFI) as non-frail (NF, score 0,1), pre-frail (PF, score 2, 3) and severe frail (SF, score >4).
Inflammatory biomarkers | preoperatively
  Upon admission and immediate before surgery upper limits of white blood cells (WBC) within normal range (WBC >8 10^3/μL), NLR (neutrophils/lymphocytes), PLR (platelets/lymphocytes), CRP (C-reactive protein) and CLR (CRP/lymphocytes), will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, Professor, Study Chair — University of Thessaly
Locations (2):
- Greece (2):
  - Larissa University Hospital, Larissa, Thessaly
  - UHL, Larissa, Thessaly